CLINICAL TRIAL: NCT03938727
Title: Cardiovascular Risk Factors, Aging and Dementia (III Follow-up)
Brief Title: Cardiovascular Risk Factors, Aging and Dementia
Acronym: CAIDE
Status: Completed | Type: Observational
Sponsor: University of Eastern Finland (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAIDE85+
Record Dates: First submitted 2019-04-04; First posted 2019-05-06 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Dementia
Keywords: Dementia; Aging; Alzheimer's Disease; Cognition; Frailty; Epidemiology; Lifestyle; Cardiovascula Risk Factors
MeSH Terms: conditions — Dementia; Alzheimer Disease; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The global challenges caused by dementia affect society from both the public health and economic perspective, and are exacerbated by the rapid growth of the population in the oldest age groups. Reducing the risk of developing dementia and improving the overall health status, psychosocial wellbeing, and the quality of life of the oldest old would bear individual and public health benefits, as well as social and economic advantages. Data from long-term longitudinal cohort studies can provide invaluable information about the factors that play a key role in healthy ageing and in the development of dementia. The aim of CAIDE 85+ is to better understand the factors that, from mid- to late-life, determine the development of cognitive disorders such as dementia, as well as the overall health status, psychosocial wellbeing and quality of life in the oldest old segment of the population.

CAIDE85+ is the third follow-up of the main Cardiovascular Risk Factors, Aging and Dementia (CAIDE) study conducted in the Kuopio and Joensuu areas in Eastern Finland. During midlife, participants were initially part of two population-based health surveys (North Karelia project and FINMONICA study) carried out between 1972 and 1987. In 1998, a random sample of 2000 individuals (aged 64-79) from these cohorts were invited to participate in a first re-examination as part of the CAIDE study. A second re-examination of this population was carried out between 2005 and 2008. Individuals who are still alive and living in the Kuopio and Joensuu areas will now be invited for a third re-examination. Participants' cognitive functioning and physical fitness will be assessed, and they will be asked questions about their health status, psychosocial wellbeing, and lifestyle. Blood samples will be also collected to investigate biomarkers that may be relevant for dementia-related diseases.

DETAILED DESCRIPTION:
The Cardiovascular Risk Factors, Aging and Dementia (CAIDE) study was initiated in 1998 with the main scope of investigating the potential role of modifiable risk and protective factors in the development of dementia. 2000 people, who, in mid-life between 1972 and 1987, had taken part in the North Karelia, and FINMONICA survey studies, were invited to participate. These previous cohort studies focused mostly on cardiovascular disease and related risk factors and provided baseline data for the CAIDE study. Within CAIDE, two follow-ups have been carried out so far, the first in 1998 and the second between 2005 and 2008, on average 21 and more than 30 years after the baseline studies, respectively.

The CAIDE study has, so far, provided essential knowledge on several midlife risk and protective factors for dementia, including interactions between genetics and lifestyle. In addition, the CAIDE Dementia Risk Score was developed as the first tool for predicting the risk of late-life dementia in middle-aged people, based on their lifestyle and cardiovascular risk profiles.

Ten years after the second re-examination, the CAIDE participants are now well in their middle 80s' or older. Despite being the fastest growing segment of the population, this age group has been only rarely the subject of similar observational studies. By investigating the health status, quality of life, and overall psycho-physical functionality in this population the investigators aim to further examine risk and protective factors for dementia. To this aim, a life-course approach will be applied on a unique longitudinal population-based dataset spanning over 40 years, a very long period of time that is rarely achievable in observational studies. The results will also provide insights on the predictors and determinants of quality of life and psychosocial wellbeing in the oldest old.

CAIDE85+ is the third follow-up of the main CAIDE study. At baseline (midlife), data on e.g. socio-demographics, lifestyle, anthropometric measurements, blood pressure, blood markers, and medical history were recorded. In addition, the first and second late-life re-examinations included cognitive assessments (three-step protocol for the diagnosis of Mild Cognitive Impairment and dementia), APOEƐ4 genotyping, and more detailed data on psychosocial factors, and medication use. In principle, the same measurements and methods will be used in CAIDE 85+, except for modifications/adaptations required by the specifics of the 85+ study population, or recent scientific developments related to the aims of the study. New developments compared with previous re-examinations include e.g. single-step assessment of cognitive status for all participants; more detailed assessment of physical functioning, multimorbidity and frailty; inclusion of questionnaires on oral health, sleep quality, malnutrition, and health-related quality of life.

Potential participants will be identified within the original CAIDE cohort, i.e. individuals who are still alive and living in the area where the study takes place (Kuopio and Joensuu, Finland).

ELIGIBILITY:
Inclusion Criteria:

* Previous invitation to the first CAIDE follow up (1998)
* Being still alive and living in the Kuopio and Joensuu areas (Finland)

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants will be selected from the original cohort of people who were invited to participate in the first CAIDE follow-up. This includes 2000 people randomly selected from the previous North Karelia and FINMONICA surverys carried out between 1972 and 1987. Any member of the original CAIDE sample still alive and living in the Kuopio or Joensuu areas (Finland) will be invited.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Cognitive performance, CERAD | One assessment within 8 weeks from consent
  Finnish version of CERAD (Consortium to Establish a Registry for Alzheimer´s Disease). Score range: 0-100, higher score indicates a better outcome.
Cognitive performance, MMSE | One assessment within 8 weeks from consent
  Mini Mental State Examination. Score range: 0-30, higher score indicates a better outcome.
Clinical Dementia Rating, units on a scale. | One assessment within 8 weeks from consent
  Influence of cognitive impairment on the ability to conduct everyday activities on six domains (memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care). Score ranges: 0-3 (individual domain), 0-18 (total score as sum of the six domains). Lower score indicates a better outcome.
Activity of Daily Living, Katz Index. | One assessment within 8 weeks from consent
  Self-reported questionnaire ranking the independence in six basic daily functions. For each activity, the participant is rated either dependent (0 points) or independent (1 point). The total score score ranges 0-6 and a higher score indicates a better outcome.
Activity of Daily Living, Lawton-Brody Scale. | One assessment within 8 weeks from consent
  Self-reported questionnaire assessing the level of functioning in eight daily activities necessary for living in the community. For each activity, the participant is rated either dependent (0 points) or independent (1 point). Score ranges 0-8 and a higher score indicates a better outcome.
Dementia and mild cognitive impairment | Through study completion, an average of 2 years
  MCI and dementia diagnoses (including type of dementia) will be ascertained from the participants' medical records. Data linkage to national registers.

SECONDARY OUTCOMES:
Multimorbidity | Through study completion, an average of 2 years
  Total number of diagnoses of concomitant chronic medical conditions ascertained based on medical history data from e.g. previous follow-up data, as well as medical records. Data linkage to national registers.
Frailty Index, units on a scale. | One assessment within 8 weeks from consent
  Fried Frailty phenotype, defined by assessing five criteria: unintentional weight loss, self-reported exhaustion, weakness by grip strength, slow walking speed, and low physical activity. One point is attributed when each of the five criteria is met. Score range: 0-5, a lower score indicates a better outcome.
Short Physical Performance Battery, units on a scale. | One assessment within 8 weeks from consent
  Physical performance is assessed in three domains: balance standing (score range: 0-4), chair standing (score range: 0-4), and gait speed (score range: 0-4). The total score (range: 0-12) is the sum of the three scores. A higher score indicates a better outcome.
Physical functioning - Hand-grip strength, kg. | One assessment within 8 weeks from consent
  The test measures the maximum isometric strength of the hand and forearm muscles and it is carried out with the aid of a hand-grip dynamometer.
Self-reported physical activity | One assessment within 8 weeks from consent
  Number of days/week in which physical activity is carried out for at least 20 minutes.
Psychosocial wellbeing - Hopelessness, units on a scale. | One assessment within 8 weeks from consent
  Self-reported questions inquiring about sense of hopelessness.
Psychosocial wellbeing - Social network | One assessment within 8 weeks from consent
  Self-reported questions inquiring about social network.
Psychosocial wellbeing - Subjective memory complaints, units on a scale. | One assessment within 8 weeks from consent
  22-item self-reported questionnaire inquiring on subjective memory. Score range: 0-66, a lower score indicates a better outcome.
Psychosocial wellbeing - Anxiety, units on a scale | One assessment within 8 weeks from consent
  State Trait Anxiety Inventory (STAI -6), self-reported 6-item questionnaire inquiring about sense of anxiety. Score range: 0-18, a lower score indicates a better outcome.
Psychosocial wellbeing - Depression, units on a scale. | One assessment within 8 weeks from consent
  Beck Depression Inventory (BDI), a 21-item self-reported questionnaire including inquiring about symptoms of depression. Score range: 0-63. A lower score indicates a better outcome.
Psychosocial wellbeing - Life events | One assessment within 8 weeks from consent
  Self-reported list of 12 significant life events.
Psychosocial wellbeing - Sleep quality, units on a scale. | One assessment within 8 weeks from consent
  Pittsburgh Sleep Quality Index (PSQI), measuring the quality and patterns of sleep in older adults. Score range 0-21. A lower score indicates a better outcome.
Oral health | One assessment within 8 weeks from consent
  Self-reported questions inquiring about oral health.
Nutritional status, units on a scale. | One assessment within 8 weeks from consent
  Mini Nutritional Assessment (MNA), a screening tool specifically designed for older adults to help identify elderly people who are malnourished or at risk of malnutrition. The assessment consists of six items evaluated by the assessor. A score (0-3 or 0-2) is attributed to each item based on the assessor's evaluation. The overall score ranges 0-14, and a higher score indicates a better outcome.
Dietary habits | One assessment within 8 weeks from consent
  Self-reported questions inquiring about dietary habits.
Health-related quality of life, units on a scale. | One assessment within 8 weeks from consent
  RAND 36-Item Health Survey 1.0, a 36-item self-reported questionnaire inquiring about health related quality of life. Score range: 0-100, a higher score indicates a better outcome.

OTHER OUTCOMES:
Blood pressure, mmHg. | One assessment within 8 weeks from consent
  Systolic and diastolic blood pressure
BMI, kg/m2 | One assessment within 8 weeks from consent
  Body mass index
Waist-hip ratio, cm. | One assessment within 8 weeks from consent
  Hip-waist Circumference: measured to nearest 0.1cm
Blood glucose, mmol/L | One assessment within 8 weeks from consent
  Fasting Glucose
Glycated hemoglobin, mmol/mol | One assessment within 8 weeks from consent
  Blood level of glycated haemoglobin A1c (HbA1c)
Cholesterol, mmol/L | One assessment within 8 weeks from consent
  Total blood cholesterol level
LDL cholesterol, mmol/L | One assessment within 8 weeks from consent
  Blood low density lipoprotein cholesterol level
HDL, mmol/L | One assessment within 8 weeks from consent
  Blood high density lipoprotein cholesterol level
Triglycerides, mmol/L | One assessment within 8 weeks from consent
  Blood triglycerides level
Creatinine, mg/dl | One assessment within 8 weeks from consent
  Blood creatinine level
CRP, mg/L | One assessment within 8 weeks from consent
  Blood C-reactive protein level
Smoking habits | One assessment within 8 weeks from consent
  Self-reported questions about smoking status: never/past/current
Current medications | One assessment within 8 weeks from consent
  Self-reported list of medication currently used
Medical history | Through study completion, an average of 2 years
  Diagnoses, hospitalizations and other relevant events related to the participants healthcare will be recorded from national registers
Sociodemographic factors | One assessment within 8 weeks from consent
  Marital status, living/domicile setting, current yearly income, work history.
Leisure activities | One assessment within 8 weeks from consent
  Self-reported questions inquiring about 12 leisure-time activities.

CONTACTS AND LOCATIONS:
Overall Officials: Miia Kivipelto, MD, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

REFERENCES:
- [Derived] Barbera M, Kulmala J, Lisko I, Pietila E, Rosenberg A, Hallikainen I, Hallikainen M, Laatikainen T, Lehtisalo J, Neuvonen E, Rusanen M, Soininen H, Tuomilehto J, Ngandu T, Solomon A, Kivipelto M. Third follow-up of the Cardiovascular Risk Factors, Aging and Dementia (CAIDE) cohort investigating determinants of cognitive, physical, and psychosocial wellbeing among the oldest old: the CAIDE85+ study protocol. BMC Geriatr. 2020 Jul 10;20(1):238. doi: 10.1186/s12877-020-01617-5. PMID 32650731